CLINICAL TRIAL: NCT04769544
Title: Comparison Between Medial Pivot Versus Symmetric Insert Total Knee Arthroplasty: A Randomized Controlled Study
Brief Title: Comparison Between Medial Pivot Versus Symmetric Insert Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elda University Hospital (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Alejandro Lizaur-Utrilla, PhD, MD, Head of Orthopaedic Surgery Department, Elda University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MedialPivotPTR2021
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Total knee arthroplasty; Medial pivot
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Patients will be treated surgically with a TKA. The two patient groups will include: 1) Study group treated a medial pivot TKA; 2) Control group treated with a conventional TKA.
  Patients will be followed at regular postoperative intervals by orthopaedic surgeons not involved in the surgeries or cares.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind. Patients will be allocated into two groups based on randomized 20-block method by an independent assistant using computer generated randomization. Both patients and evaluators will be blinded with regard to the TKA design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial pivot group (Active Comparator): Device used: medial pivot total knee arthroplasty design
  Interventions: Device: total knee arthroplasty with medial pivot tibial insert or symmetrical insert
- Conventional group (Active Comparator): Device used: conventional total knee arthroplasty design
  Interventions: Device: total knee arthroplasty with medial pivot tibial insert or symmetrical insert

INTERVENTIONS:
Device: total knee arthroplasty with medial pivot tibial insert or symmetrical insert — standard surgical implantation of total knee arthroplasty

SUMMARY:
The functional outcome and longevity of total knee arthroplasty (TKA) is still a concern. Despite various developments in TKA designs, including fixed or mobile bearing, cruciate retaining or posterior stabilized, multi or single radius, it remains unclear which design is superior for achieving a physiological kinematic.

In normal healthy knees the medial and lateral tibial condyles are different: the medial is almost flat while the lateral is somewhat convex. Thus, the movement during flexion is asymmetric: during the flexion, the medial condyle is stable throughout the range of motion while the lateral condyle slides anteroposteriorly with respect to femur). Therefore, the native knee requires a specific degree of rollback of the lateral compartment coupled with a medial pivot, which leads to an external axial rotation of the femur. This rollback is thought to be even more pronounced with increasing knee flexion angles to enable deep flexion without excessive shear forces acting at the patella or overloading the extensor mechanism.

In addition, stability throughout flexion is a crucial element to normal knee function. Most TKA designs removal of the ACL, and the PCL in posterior-stabilized design, but the TKA do not fully restore the function of those ligaments.

Based on this philosophy, the medial pivot TKA was designed to provide better function, patient satisfaction and increased survival.

The objective of this study is to analyze whether the medial pivot design provides better outcome and prosthesis survival than conventional total knee arthroplasty.

DETAILED DESCRIPTION:
Candidates for the study will be consecutive patients eligible for total knee arthroplasty (TKA) at our center. All patients meeting inclusion criteria will be recruited for enrollment into the study. Informed consent will be obtained from the patient prior to randomization.

At that time, each patient will be randomized into one of two groups by an independent staff using computer generated randomization and allocation concealment. The two patient groups will include:

1. Study group: patients treated with a medial pivot TKA.
2. Control group: patients treated with a conventional TKA. Patients will be preoperatively assessed and postoperatively at regular intervals (6mo, 12 mo, and then annually) by orthopaedic surgeons not involved in the surgeries or cares.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee
* 50 years and older
* Participants must be able to give informed consent

Exclusion Criteria:

* Inflammatory arthritis
* Traumatic etiology
* Neurologic disease
* Neoplastic disease
* Morbid obesity
* Severe collateral ligament instability (> 10° varus/valgus)
* Severe knee misalignment (greater than 10° of varus or valgus)
* Flexion contracture greater than 15º
* Prior surgery on the affected knee (except meniscus)
* Knee arthroplasty in the contralateral knee

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Knee Society Score | 2 years
  Functional KSS score (range 0-100) with higher scores as better outcome. A good result is defined as 70 points or greater

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Lizaur-Utrilla, MD, PhD, Principal Investigator — Elda University Hospital
Locations (1):
- Elda University Hospital, Elda, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Request to the principal investigator